CLINICAL TRIAL: NCT03335657
Title: Improving Recovery After Orthopaedic Trauma: Cognitive-Behavioral Based Physical Therapy (CBPT)
Acronym: CBPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W81XWH-16-2-0060
Record Dates: First submitted 2017-10-25; First posted 2017-11-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Lower Extremity Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBPT Treatment (Experimental): The CBPT intervention delivers a patient-oriented cognitive-behavioral self-management program to improve physical function and reduce pain, through reductions in pain catastrophizing and fear of movement and increases in self-efficacy. The program consists of six weekly telephone sessions with a trained physical therapist. Sessions cover an introduction and rationale for treatment in addition to techniques such as deep breathing, graded activity plan and goal-setting, distraction techniques, automatic thoughts, coping self-statements, being present-minded, and relapse prevention and symptom management plans. At the end of the 6th week, patients will build individualized recovery plans with selected strategies and details on frequency of practice.
  Interventions: Other: CBPT
- Education Treatment (Placebo Comparator): The education program provides a postoperative recovery and is based on education that would typically be provided by a treating physician or a physical therapist in an outpatient setting. The education program is matched to the CBPT treatment in terms of session frequency and contact with the study therapist. The therapist will call weekly to check in with the patient and encourage him/her to read the manual. Manuals contain educational information on injury patterns and symptoms, stress and recovery, benefits of physical therapy, and importance of daily exercise, and ways to promote healing. Education on sleep hygiene, energy management, healthy eating, and preventing future injury are also provided.
  Interventions: Other: Education Treatment

INTERVENTIONS:
Other: CBPT — The CBPT program focuses on a patient-oriented cognitive-behavioral self-management approach to improve physical function and reduce pain, through reductions in pain catastrophizing and fear of movement and increases in self-efficacy.
  Arms: CBPT Treatment
Other: Education Treatment — Participants receiving the education control arm are receiving a placebo intervention to control for the attention of the interventionist. They will receive standardized educational material addressing recovery from orthopaedic trauma.
  Arms: Education Treatment

SUMMARY:
The goal of the CBPT study is to determine the efficacy of the CBPT program for improving outcomes in service members and civilians at-risk for poor outcomes following traumatic lower-extremity injury. Primary outcome is physical function measured through a patient-reported questionnaire and physical performance tests. Secondary outcomes include pain and general health. Tertiary outcome is return to work/duty.

DETAILED DESCRIPTION:
Following extremity injury, referral (and direct access) to physical therapy (PT) is considered standard of care. And, while PT strategies are commonly impairment focused, clinicians across multiple subspecialties of physical therapy recognize the importance of addressing pain and pain-related psychosocial factors as strong predictors of chronic pain as well as long-term physical and psychological disability.

Cognitive-behavioral therapy (CBT) interventions have documented positive influence on psychosocial factors in patients with chronic pain. CBT-based self-management programs have also demonstrated improvement in patient outcomes and the adoption of a physically active lifestyle, as well as improvement in fear-avoidance beliefs and self-efficacy, in various populations with chronic conditions. These evidence-based CBT and self-management strategies provide the basis for the study intervention.

The proposed project will conduct a multi-center, randomized controlled trial to determine the efficacy of the CBPT program in patients at-risk for poor outcomes following traumatic lower-extremity injury. Central hypothesis is that delivery of CBPT by physical therapists over the telephone will improve outcomes, through reductions in pain catastrophizing and fear of movement and improvement in pain self-efficacy. The investigators propose a large, rigorous evaluation of the CBPT program in patients with lower extremity trauma with the goal of engaging civilians and service members in their own care and improving pain and functional outcomes.

Specific Aim 1 To determine the efficacy of the CBPT program for improving outcomes in service members and civilians at-risk for poor outcomes following traumatic lower-extremity injury. Primary outcome is physical function measured through a patient-reported questionnaire. Secondary outcomes include physical performance tests, pain and general health. Tertiary outcome is return to work/duty.

Specific Aim 2 To determine whether changes in the intermediary outcomes of pain catastrophizing, fear of movement, and self-efficacy at 6 months are associated with improvement in outcomes 12 months after hospital discharge.

Specific Aim 3 To determine whether subgroups of patients are more likely to benefit from the CBPT program.

Specific Aim 4 To examine the value of CBPT relative to Education using Markov decision-analysis.

ELIGIBILITY:
Inclusion criteria:

1. Ages 18-60 yrs inclusive
2. Patients with at least one acute orthopaedic injury to the lower extremities or pelvis/acetabulum (determination based on information available at the time of enrollment).
3. Injury resulting from a moderate to high energy force (e.g. motor vehicle or motorcycle crash, fall > 10 ft, gun shot, blunt trauma)
4. Patients receiving operative fixation for one or more acute orthopaedic injuries at a participating hospital. Patients should be recruited at the time of primary injury, not revision or complication surgery
5. Presence of psychosocial risk factors for poor outcomes (defined as a score greater than 30 on the Pain Catastrophizing Scale (PCS) or a score equal to or greater than 39 on the Tampa Scale for Kinesiophobia (TSK) or a score equal to or less than 40 on the Pain Self Efficacy Scale (PSES)). These risk factors will be identified between 2 and 8 weeks after hospital discharge.

Exclusion criteria:

1. Non-English speaking
2. Patients who are unable to start the program within 12 weeks of discharge from hospital because of multiple readmission, admission to a rehabilitation facility, or other extenuating circumstances
3. Patients with moderate or severe traumatic brain injury (TBI), as evidenced by intracranial hemorrhage present on admission CT. If no CT performed, patient assumed not to have moderate or severe TBI
4. Patients with major amputations of the upper or lower extremities (great toe, thumb, or proximal to the wrist or ankle)
5. Patients who require a Legally Authorized Representative (as defined by an inability to answer the "Evaluation of Give Consent" questions)
6. Patients non-ambulatory pre-injury or due to an associated spinal cord injury
7. History of dementia or Alzheimer's disease based on medical record or patient self-report
8. History of neurological disorder, disease or event, resulting in prior cognitive and/or physical impairment, such as prior TBI or stroke based on medical record or patient self-report
9. Presence of schizophrenia or other psychotic disorder based on medical record or patient self-report
10. Current alcohol and/or drug addiction based on medical record or patient self-report
11. Severe problems with maintaining follow-up expected (e.g. patients who are incarcerated or homeless)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 633 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Physical Function- self-reported capability to carry out activities | 12 months
  Physical Function measured through Patient Reported Outcome Measurement Information System (PROMIS)/ Physical Function (short form) domain to assess one's ability to carry out activities that require a combination of skills, often within a social context. This instrument has five response options ranging in value from one to five for each question. The total raw score is the sum of values of the response for each question The highest possible raw score is 40 which represents the worse outcome. The lowest possible score is 8 and it represents the better outcome.

SECONDARY OUTCOMES:
Pain_ self reported | 12 months
  Pain measured through Patient Reported Outcome Measurement Information System (PROMIS)/ Pain Intensity (short form) Domain at 12-months following hospital discharge. This tool has five response options ranging in value from one to five for each question. The total raw score is the sum of values of the response for each question The highest possible raw score is 15 which represents the worse outcome. The lowest possible score is 3 and it represents the better outcome.
General Health | 12 months
  General Health measured through the Veterans RAND 12 Item Health Survey (VR-12)/ General Health Domain at 12-months following hospital discharge. This instrument has five response options ranging in value from one to five for each question. The total raw score is the sum of the values of the responses for each question. The highest possible raw score is 60, which represents the better outcome. The lowest possible score is 12, and it represents the worse outcome.
Physical Function- Balance and Agility | 12 months
  Balance and Agility measured through the Four Square Step test. Each individual will have time scores based on performance. Higher scores represent worse outcomes.
Physical Function- Mobility and Power | 12 months
  Mobility and Power measured through the Timed Stair Ascent test. Each individual will have time scores based on performance. Higher scores represent worse outcomes.
Physical Function-Leg Strength, Endurance, and Mobility | 12 months
  Leg Strength, Endurance, and Mobility measured through the Sit to Stand Five Times
Physical Function- Gait Speed | 12 months
  Gait Speed measured through 10-Meter Walk test. Each individual will have time scores

OTHER OUTCOMES:
Return to work/duty | 6 months
  Measured through the rate of return to work/duty 6 months post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Swygert, PhD, Principal Investigator — Vanderbilt University Medical Center; Katherine Frey, PhD, Study Director — Johns Hopkins University
Locations (8):
- United States (8):
  - Florida Orthopaedic Institute, Tampa, Florida
  - Methodist Hospital, Indianapolis, Indiana
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Carolinas Medical Center, Charlotte, North Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Archer KR, Davidson CA, Alkhoury D, Vanston SW, Moore TL, Deluca A, Betz JF, Thompson RE, Obremskey WT, Slobogean GP, Melton DH, Wilken JM, Karunakar MA, Rivera JC, Mir HR, McKinley TO, Frey KP, Castillo RC, Wegener ST; METRC. Cognitive-Behavioral-Based Physical Therapy for Improving Recovery After Traumatic Orthopaedic Lower Extremity Injury (CBPT-Trauma). J Orthop Trauma. 2022 Jan 1;36(Suppl 1):S1-S7. doi: 10.1097/BOT.0000000000002283. PMID 34924512